CLINICAL TRIAL: NCT06736288
Title: Randomized, Double Blind, Placebo Controlled, Two-Arms, Multicenter, Post Authorization Efficacy and Safety Study (PAES) to Confirm and Collect More Clinical Data of Buccalin® Tablets In the Prophylaxis of Recurrent Lower Respiratory Tract Infections (RLRTIs).
Brief Title: Post Authorization Efficacy and Safety Study (PAES) to Confirm and Collect More Clinical Data of Buccalin® Tablets In the Prophylaxis of Recurrent Lower Respiratory Tract Infections (RLRTIs).
Acronym: BUC-01-23
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorio Farmaceutico SIT srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BUC-01-23; 2024-512937-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Infection; Lower Respiratory Tract Infection (LRTI)
MeSH Terms: conditions — Respiratory Tract Infections | interventions — buccalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUCCALIN® gastro-resistant tablets (Active Comparator): mixture of Streptococcus pneumoniae I, II, III, Streptococcus agalactiae, Staphylococcus aureus, Haemophilus influenzae
  Interventions: Drug: BUCCALIN®
- Placebo (Placebo Comparator): gastro-resistant tablets containing only excipients
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BUCCALIN® — Gastro-resistant tablets (mixture of Streptococcus pneumoniae I, II, III, Streptococcus agalactiae, Staphylococcus aureus, Haemophilus influenzae).
  The recommended dosage is 1 tablet on day 1, 2 tablets on day 2, and 4 tablets on day 3 and should be taken in the morning on an empty stomach.
  Arms: BUCCALIN® gastro-resistant tablets
Other: Placebo — Gastro-resistant tablets containing only excipients). The recommended dosage is 1 tablet on day 1, 2 tablets on day 2, and 4 tablets on day 3 and should be taken in the morning on an empty stomach.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess if BUCCALIN® works In the Prophylaxis of Recurrent Lower Respiratory Tract Infections (RLRTIS). It will also evaluate the safety of BUCCALIN®.

The primary aim is to reduce the number of infection episodes in the treatment period (12 months) in the BUCCALIN® group versus the Placebo group.

Patients diagnosed with RLRTIS will be screened for enrolment. Patients will be requested to provide informed consent before the start of the study related assessments.

Eligible patients who meet the study inclusion and exclusion criteria will be randomized with a 1:1 ratio allocation to the 2 treatment groups.

Researchers will compare BUCCALIN® (gastro-resistant tablets) to a placebo (gastro-resistant tablets containing only excipients) to treat RLRTIS.

Patients who participate in the study will perform several study visits divided as reported below:

* Run-in phase (12 months): patients will not receive any treatment. This phase is designed to increase adherence to the study and reduce loss to follow-up in the clinical trial. During this phase, patients should experience ≥ 2 episodes of RTIs to be eligible for the Treatment period.
* Treatment period (12 months): patients will receive BUCCALIN® or Placebo treatment for 12 consecutive months (3 days per month, posology as per authorized SmPC).
* Follow-up period (12 months): patients will not receive any treatment. This phase is designed to observe how patients respond to treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and able to provide voluntary informed consent and to follow protocol requirements.
2. Male or females from 18 to 99 years old, (Adult, Older Adult).
3. Patients with Recurrent LRTIs including tracheitis, tracheobronchitis, acute bronchitis and exacerbations of chronic lung disease (asthma and/or COPD and/or bronchiectasis), who present with both of the following:

   a) ≥2 episodes within 12 months prior to the run-in period based on patient reported medical history (to access the run-in period) b) ≥2 episodes during the run-in period documented by appropriate microbiological diagnostic test (to access the treatment period)
4. Patients:

   1. not vaccinated or
   2. vaccinated against the most common pathogens for respiratory infectioan (within 12 months prior to the run-in period or during the run-in period, but not during the treatment period)*:

      - Anti-pertussis vaccination

      - Covid-19 vaccination

      - Respiratory Syncytial Virus vaccination

      - Influenza vaccination

      - Pneumococcal vaccination

      * Patients vaccinated with other types of vaccines that have no effect on the lower respiratory tract (e.g. hepatitis b vaccination, shingles/herpes zoster vaccination, papilloma virus vaccine), in addition to the ones listed above, may also be included.

Exclusion Criteria:

RUN-IN period

1. Female patient: pregnant, lactating or planning pregnancy (Female of child-bearing potential will undergo urine pregnancy test).
2. Female of potential child-bearing that does not use at least one effective contraceptive method for the entire study.
3. Contraindication or known hypersensitivity to the active ingredients of bacterial lysates or any excipients listed in the ingredients.
4. Pneumonia (based on the EMA Referral Procedure EMEA/H/A-31/1465).
5. Known history of tuberculosis and/or cystic fibrosis.
6. Known history of immunodeficiency diseases (e.g., HIV infection, AIDS, or any type of congenital or iatrogenic immune deficiency, including IgA deficiency).
7. Severe heart failure (NYHA class III and IV).
8. Haematologic diseases including severe anaemia (defined according to the National Cancer Institute as Hemoglobin < 8.0 g/dL).
9. Renal failure (eGFR < 30 mL/min).
10. History of known liver damages defined by the METAVIR classification (F1-F4)*.
11. Malignancies with a remission period of < 5 years.
12. Wheezing documented to be caused by gastroesophageal reflux**.
13. Patient legally or mentally incapacitated unable to give informed consent for the participation in this study.
14. Patient who is unable or unwilling to comply with the appointments or with all the requirements of the Protocol.
15. History of autoimmune diseases and acute intestinal infections, as reported in Buccalin® SmPC.

    * This criterion only applies to patients with known liver disease who can produce valid fibroscan and/or biopsy results and bring them for demonstration.

      * The criterion can only be applied if the patient presents clinically reliable documentation that the wheezing is not due to a lung disease (i.e. gastroscopy).

TREATMENT period

1. Female patient: pregnant, lactating or planning pregnancy (Female of child-bearing potential will undergo urine pregnancy test).
2. Female of potential child-bearing that does not use at least one effective contraceptive method for the entire study.
3. Contraindication or known hypersensitivity to the active ingredients of bacterial lysates or any excipients listed in the ingredients.
4. Pneumonia (based on the EMA Referral Procedure EMEA/H/A-31/1465).
5. Known history of tuberculosis and/or cystic fibrosis.
6. Known history of immunodeficiency diseases (e.g., HIV infection, AIDS, or any type of congenital or iatrogenic immune deficiency, including IgA deficiency).
7. Severe heart failure (NYHA class III and IV).
8. Haematologic diseases including severe anaemia (defined according to the National Cancer Institute Hemoglobin < 8.0 g/dL).
9. Renal failure (eGFR < 30 mL/min).
10. History of known liver damages defined by the METAVIR classification (F1-F4)*.
11. Malignancies with a remission period of < 5 years.
12. Injection or oral administration of steroids within 4 weeks prior to randomization**.
13. Use of immunosuppressants, immunostimulants, or gamma globulins within 6 months prior to randomization.
14. Previous use within 6 months prior to randomization or ongoing use of bacterial lysates.
15. Any major surgery within the last 3 months prior to randomization.
16. Wheezing documented to be caused by gastroesophageal reflux***.
17. Patient legally or mentally incapacitated unable to give informed consent for the participation in this study.
18. Patient who is unable or unwilling to comply with the appointments or with all the requirements of the Protocol.
19. History of autoimmune diseases and acute intestinal infections, as reported in Buccalin® SmPC.

    * This criterion only applies to patients with known liver disease who can produce valid fibroscan and/or biopsy results and bring them for demonstration.

      * In these instances, patients may undergo a washout period of 4 weeks to qualify for the treatment period.

        * The criterion can only be applied if the patient presents clinically reliable documentation that the wheezing is not due to a lung disease (i.e. gastroscopy).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
RLRTIs Episodes: Reduction in the number of infection episodes in the treatment period (12 months) in the Buccalin® group versus the Placebo group. | From the enrollment to the end of the treatment at 24 months

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (9):
  - AOU Ss. Antonio E Biagio E C.Arrigo, Alessandria
  - AOU Policlinico G. Rodolico-San Marco, Catania
  - ASST Fatebenefratelli Sacco, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST Santi Paolo e Carlo, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Humanitas Mirasole S.p.A, Milan
  - AOU Policlinico Tor Vergata, Roma
  - AOU di Sassari, Sassari
- University clinic for infectious diseases and febrile conditions, Medical Faculty, Ss Cyril and Methodius University, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No